CLINICAL TRIAL: NCT02746328
Title: Add-on Study for Protocol G200802 (NCT02463032): Effect of GTx-024 on Maximal Neuromuscular Function and Lean Body Mass
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigational drug development was halted.
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G200802a
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: ER+ and AR+ Breast Cancer
MeSH Terms: interventions — ostarine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GTx-024 9 or 18 mg (Experimental): Patients enrolled in G200802 receiving GTx-024 9 or 18 mg
  Interventions: Drug: GTx-024 9 or 18 mg

INTERVENTIONS:
Drug: GTx-024 9 or 18 mg — Patients enrolled in G200802 receiving GTx-024 9 or 18 mg
  Other Names: Enobosarm

SUMMARY:
This is a multiple site, proof of concept feasibility study to describe the effect of GTx-024 9 or 18 mg on physical function in female subjects, from protocol G200802, with ER+/AR+ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. In screening for, and ultimately randomized into, protocol G200802
2. Give voluntary, written and signed, informed consent for this add-on study
3. Age 18 to 70 years old
4. Physically capable of mounting and riding a stationary bicycle
5. Subject agrees to not significantly alter physical activity or current physical training during the study period

Exclusion Criteria:

1. Subject has a concomitant medical condition that precludes adequate study treatment compliance or assessment, or increases subject risk, in the opinion of the Investigator
2. Subjects unwilling to or unable to comply with the protocol
3. Any other condition which per investigators' judgement may increase subject risk

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Maximal Power Production | 24 Weeks
  Describe the effect of 24 weeks of treatment of GTx-024 on maximal power production as assessed by inertial-load cycle ergometry

SECONDARY OUTCOMES:
Maximal Power Production | 12 Weeks
  Describe the effect of 12 weeks of treatment of GTx-024 on maximal power production as assessed by inertial-load cycle ergometry
Lean Body Mass | 24 Weeks
  Describe the effect of 24 weeks of treatment of GTx-024 on lean body mass (LBM) as assessed by CT images of the lumbar region from L3 to the iliac crest
Lean Body Mass | 12 Weeks
  Describe the effect of 12 weeks of treatment of GTx-024 on LBM as assessed by CT images of the lumbar region from L3 to the iliac crest
Maximal Power Production, Scaled to Total Body Mass | 24 Weeks
  Describe the effect of 24 weeks of treatment of GTx-024 on maximal power production scaled (Watts/kilogram) to total body mass (TBM), as assessed by inertial-load cycle ergometry
Maximal Power Production, Scaled to Lean Body Mass | 24 Weeks
  Describe the effect of 24 weeks of treatment of GTx-024 on maximal power production scaled (Watts/kilogram) to LBM, as assessed by inertial-load cycle ergometry
Optimal Pedaling Rate | 24 Weeks
  Describe the effect of 24 weeks of treatment of GTx-024 on optimal pedaling rate

OTHER OUTCOMES:
Exploratory Objective | 24 Weeks
  Describe the impact of baseline measures and measures obtained throughout the study on maximal power production and its change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hannah M Linden, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, School of Medicine, Seattle, Washington, United States